CLINICAL TRIAL: NCT01930760
Title: Supporting Physicians With Education And Know-how in Identifying and Motivating Overweight Kids: SPEAK IM OK
Brief Title: Supporting Physicians With Education And Know-how in Identifying and Motivating Overweight Kids
Acronym: SPEAK IM OK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000013526
Record Dates: First submitted 2013-08-25; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Obesity
Keywords: pediatric; Childhood Obesity; motivational interviewing; pediatric primary care physicians
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational Intervention Group (Experimental)
  Interventions: Behavioral: Standard Medical Training Educational
- Behavioural Intervention Group (Experimental)
  Interventions: Behavioral: Motivational Interviewing behavioural

INTERVENTIONS:
Behavioral: Standard Medical Training Educational — Educational is modeled on the Theory of Planned Action, which proposes that unless people believe that their actions can have an effect on the desired outcome they have little incentive to act or persevere in the face of difficulties. Based on this theory we will be providing physicians with information on how to calculate, plot and track BMI and how this can be associated with identification of overweight children before they present with symptoms of obesity. This intervention will attempt to demonstrate that BMI calculating, plotting and tracking are useful diagnostic monitoring tools and that their actions may lead to more effective prevention and/or treatment.
  The education intervention will not prescribe specific discussion initiation tools, although the participants will not be prevented from independently changing their communication behaviour.
  Arms: Educational Intervention Group
Behavioral: Motivational Interviewing behavioural — The behavioural intervention will incorporate specific Motivational Interviewing (MI) tools and information from a previously completed qualitative study with obese children (Obadia et al.). This study generated suggestions of how physicians can encourage children to think positively about making changes towards a healthier body weight. This intervention is designed to address physicians' lack of self-efficacy in communicating with children and their families about achieving a healthy body weight, and therefore would likely benefit from the input from children and the patient-centred theme of MI. It is based on the Trans-Theoretical Model and Stages of Change which postulates that people follow a step-wise progression towards change with specific constructs that need to be addressed before moving to the next step. These constructs are integral to the principles of MI
  Arms: Behavioural Intervention Group

SUMMARY:
The proposed study is a randomized control trial evaluating the efficacy of two training programs in increasing physician identification, documentation, and motivation of overweight children. Pediatric primary care physicians will be recruited from the College of Physician and Surgeons of Ontario and randomized into two practice-based interventions (behavioural/educational) which are a one-time training attendance. The educational intervention will focus on the medical management of pediatric obesity, the use of Body Mass Index charts, and information about how obese children would like to be approached by their physicians. The behavioural intervention will incorporate Motivational Interviewing tools in addition to an abbreviated training program received by the educational intervention group.

DETAILED DESCRIPTION:
There are no prospective, randomized clinical studies on training physicians to effectively manage pediatric obesity using both Motivational Interviewing (MI) tools and advice from overweight children. A novel aspect of this study is that the skills taught during the trainings are made so that physician can easily incorporate them into their busy practice. The generated findings from focus groups with obese children, merged guidelines for the medical management of childhood obesity, and training in specific MI tools, also make this study unique. Primary Objective:

To determine which of two interventions (behavioural/education) is most effective in increasing discussion initiation around weight with overweight children by calculating, plotting, and tracking BMI, and increasing self-reported efficacy in counseling overweight pediatric patients. HYPOTHESIS: The behaviour change intervention will be most effective because it will achieve greater changes in the above mentioned behaviours that are maintained for 6 to 12 months. These outcomes will be influenced by counselling efficacy, frequency, and type of reported barriers and not physician demographics.

Secondary Objectives:

To evaluate current physician practices of BMI calculating, plotting and/or tracking, and discussion initiation with overweight pediatric patients, and the factors that influence these behaviours. HYPOTHESIS: Physicians do not consistently calculate, plot, and/or track BMI and/or discuss weight with their pediatric patients. These practices will be primarily influenced by physicians' characteristics, counselling efficacy, frequency and type of reported barriers

ELIGIBILITY:
Inclusion Criteria:

1. Toronto area pediatricians and family physicians who are members of the College of Physicians and Surgeons of Ontario
2. Available to attend workshop at the Hospital for Sick Children
3. Pediatric patient population of at least 25% (office audit to be completed by office staff) (to ensure sufficient contact with children and their families
4. No sub-specialty practice in obesity or related co-morbidities (This study is aimed at changing communication in primary care offices for well-child patient visits)

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in physician practice from baseline | 1 year
  Recording the changes compared to baseline for physician's practice with their overweight patients (ie calculating, plotting, and tracking BMI as well as initiate discussion around obesity)

SECONDARY OUTCOMES:
Physician Self Efficacy | Baseline, 6 and 12months after intervention
  Physicians will be asked to complete a self-efficacy questionnaire about their perception of their own abilities to initiate discussion with pediatric patients and/or their families about overweight, tendencies of frequency of BMI calculating, plotting, and tracking, identify obesity or overweight in their pediatric patients, as well as identify the type of barriers they have in preventing/treating obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Brian W McCrindle, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada